CLINICAL TRIAL: NCT02554422
Title: Messung Der Beweglichkeit Der Gehörknöchelchenkette während Einer Ohroperation. ("Objective Measurements of Ossicular Chain Mobility Using a Palpating Instrument Intraoperatively")
Brief Title: Objective Measurement of Ossicular Chain Mobility Using a Palpating Instrument Intraoperatively
Acronym: PalpEar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensoptic SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-MD-0014
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Disorder of Middle Ear; Otosclerosis of Middle Ear; Cholesteatoma, Middle Ear
MeSH Terms: conditions — Cholesteatoma, Middle Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PalpEar (Experimental): Intraoperative palpation of the ossicles using the PalpEar device, to measure mobility of the ossicle chain.
  Interventions: Device: PalpEar

INTERVENTIONS:
Device: PalpEar — Palpation of the middle-ear ossicles using the PalpEar device, to measure mobility of the ossicle chain

SUMMARY:
Feasibility of the objective measurement of the ossicular chain mobility, by using a force-measuring device based on a fiber optics sensors (PalpEar).

DETAILED DESCRIPTION:
The aim of this study was to develop and test a palpating instrument, which enables the experienced and occasional otologic surgeon to record force in three dimensions during his standard palpation of each ossicle at surgery and al-lows correlation of his subjective impression with objective measurement results. The first task was to incorporate force sensing capability into a standard 45° angulated 2.5 mm hook, which is commonly used to palpate, disconnect and luxate ossicles during middle ear surgery.

ELIGIBILITY:
Inclusion criteria:

* Adult subjects
* Normally scheduled for middle-ear or internal-ear surgery as a result of an ear disease and for whom a routine assessment of the mobility of the ossicle chain is in order.

The targeted subject population consists of patients undergoing stapedotomy for otosclerosis and subjects with a normal ossicular chain who are subject to the placement of a cochlear implant to treat hearing loss.

Exclusion criteria:

* Children
* Subjects in whom the ossicle chain is missing or incomplete
* Missing informed consent form
* Incapacitated subjects or subjects with impaired judgment capability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Measurement of the ossicle mobility through the palpation force | 1 day. The measurements are performed during day 1, in parallel with the underlying surgery, and therefore assessed within the time frame of 1 day.
  The palpation forces needed to move the middle-ear ossicles out from their resting position will be measured through a force sensing device. The measured palpation forces are measured in equivalent gram-force [gF]. The primary outcome of the study is to demonstrate if a relation can be established between the subjective feeling of the surgeon and an objective measurement of the palpation force.

SECONDARY OUTCOMES:
Difference between normal and impaired ossicular chains | 1 day. The measurements are performed during day 1, in parallel with the underlying surgery, and therefore assessed within the time frame of 1 day.
  A comparison between ossicular chains judged as "normal" by the surgeon and impaired ossicular chains will be performed, to assess if a significant difference can be extracted from the measurement of the palpation force. This would help in a future diagnosis assisted by a force sensing device.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Linder, Prof. MD, Principal Investigator — Luzerner Kantonsspital

REFERENCES:
- [Background] Huber A, Linder T, Ferrazzini M, Schmid S, Dillier N, Stoeckli S, Fisch U. Intraoperative assessment of stapes movement. Ann Otol Rhinol Laryngol. 2001 Jan;110(1):31-5. doi: 10.1177/000348940111000106. PMID 11201805
- [Background] Zöllner F. Die bisherigen Ergebnisse der Schallsondenunersuchungen. Arch Ohren-, Nasen- und Kehlkopfheilkunde 1951;159:358-364
- [Background] Shea MC Jr. Postinflammatory osteogenic fixation of the stapes. Laryngoscope. 1977 Dec;87(12):2056-65. doi: 10.1288/00005537-197712000-00012. PMID 926970
- [Background] Lau HH, Michler H, Zollner F. Versuch einer technischen Verbesserung der Schallsonde. Acta Otolaryngol 1963;56:421-7
- [Background] Gyo K, Sato H, Yumoto E, Yanagihara N. Assessment of stapes mobility by use of a newly developed piezoelectric ceramic device. A preliminary experiment in dogs. Ann Otol Rhinol Laryngol. 2000 May;109(5):473-7. doi: 10.1177/000348940010900506. PMID 10823476
- [Background] Zahnert T, Huttenbrink KB, Bornitz M, Hofmann G. [Intraoperative measurement of stapes mobility using a hand-guided electromagnetic probe]. Laryngorhinootologie. 2001 Feb;80(2):71-7. doi: 10.1055/s-2001-11896. German. PMID 11253568
- [Background] Koike T, Murakoshi M, Hamanishi S, Yuasa Y, Yuasa R, Kobayashi T, Wada H. An apparatus for diagnosis of ossicular chain mobility in humans. Int J Audiol. 2006 Feb;45(2):121-8. doi: 10.1080/14992020500377899. PMID 16566250
- [Background] Hato N, Kohno H, Okada M, Hakuba N, Gyo K, Iwakura T, Tateno M. A new tool for testing ossicular mobility during middle ear surgery: preliminary report of four cases. Otol Neurotol. 2006 Aug;27(5):592-5. doi: 10.1097/01.mao.0000226298.36327.3d. PMID 16868506
- [Background] Seidman MD, Standring RT, Ahsan S, Marzo S, Shohet J, Lumley C, Verzal K. Normative data of incus and stapes displacement during middle ear surgery using laser Doppler vibrometry. Otol Neurotol. 2013 Dec;34(9):1719-24. doi: 10.1097/MAO.0b013e3182976528. PMID 23928515
- [Background] Hato N, Stenfelt S, Goode RL. Three-dimensional stapes footplate motion in human temporal bones. Audiol Neurootol. 2003 May-Jun;8(3):140-52. doi: 10.1159/000069475. PMID 12679625